CLINICAL TRIAL: NCT01773551
Title: Development of a Quantitative Tissue Optical Index of Breast Density
Brief Title: Development of a Quantitative Tissue Optical Index of Breast Density For Prediction of Hormone Therapy Response
Status: Withdrawn | Type: Observational
Why Stopped: Not NIH defined clinical trial study
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Francisco (Other); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Thomas O'Sullivan, Ph.D.Director, Diffuse Optical Spectroscopy & Imaging Laboratory, University of California, Irvine
Other Study IDs: 20128714
Record Dates: First submitted 2013-01-14; First posted 2013-01-23 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Accessory; Breast Tissue
MeSH Terms: interventions — Breast Density

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optical Index of Breast Density: Breast Density
  Interventions: Other: Breast Density

INTERVENTIONS:
Other: Breast Density — Development of a Quantitative Tissue Optical Index of Breast Density

SUMMARY:
The purpose of this research study is to investigate whether breast density measured by a safe, painless imaging method (called Diffuse Optical Spectroscopic Imaging - DOSI) can detect the decrease of breast density in subjects who receive tamoxifen when compared to patients who do not receive any drug. If decreased density can be reliably detected, it may help determine which subjects will benefit by taking tamoxifen or other chemoprevention drugs.

DETAILED DESCRIPTION:
The goal of this study is to develop a safe, painless imaging method to measure the change in breast density caused by hormonal chemotherapy treatments such as tamoxifen. For many patients with breast cancer, chemoprevention drugs (such as tamoxifen) can reduce the risk of recurrence. However, tamoxifen can also cause serious side effects such as blood clots and an increased risk of uterine cancer. Patients would benefit from an individualized method of determining whether the chemoprevention is working. Recent studies have shown that a course of tamoxifen is more effective at reducing risk in women who exhibit >10% reduction in breast density compared to women who had little or no density change. The study suggests that breast density is a predictor of the effectiveness of tamoxifen. We propose to use an imaging method that uses safe visible and near-infrared light to measure breast tissue called diffuse optical spectroscopic imaging. Diffuse optical spectroscopic imaging allows patients to be followed through treatment with a cost-effective, bedside, handheld scanning probe. In this study, we will examine whether diffuse optical spectroscopic imaging is sensitive to the density changes induced by tamoxifen as a preventative hormonal chemotherapy agent. MRI will be used as the standard for comparison. We expect to discover that after 12-18 months, women on tamoxifen treatment will show a significant reduction in breast density compared to women not taking tamoxifen, and this change can be monitored using DOSI alone. If validated, our method could be used to determine if tamoxifen treatment is working in an individual patient and could guide doctors about the decision to end and/or switch to a different treatment. In addition, a validated index of density that can be obtained using an inexpensive, risk-free bedside technology could be applied to the challenging problem of measuring individual risk of breast cancer in the broader population.

ELIGIBILITY:
Treatment Group Inclusion Requirements

1. Premenopausal or peri-menopausal female older than 21 years of age
2. Elect to undergo, but have not yet started tamoxifen therapy;
3. Not pregnant and willing to use adequate contraception for the duration of study participation; and
4. Willing to avoid oral contraception use (which is not recommended while on tamoxifen treatment) for the duration of the study participation.

Normal Group Inclusion Requirements

1. Premenopausal or peri-menopausal female older than 21 years of age
2. Not pregnant and willing to use adequate contraception for the duration of study participation;

Exclusion (both groups) Requirements

1. Had or plan to receive any chemotherapy;
2. Have bilateral breast cancer
3. Previous treatment (chemotherapy, radiation, or surgery) to both breasts, including hormone therapy;
4. Are pregnant or nursing;
5. Have implanted prosthetic heart valves, pacemaker, neuro-stimulation devices, surgical clips (hemostatic clips) or other metallic implants;
6. Have engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or have imbedded metal fragments from military activities;
7. Have received orthodontic work involving ferromagnetic materials;
8. Are claustrophobic; or
9. Medically unstable.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups of subjects will be recruited:
  1. Pre-menopausal women who will receive the chemoprevention drug tamoxifen (treated)
  2. Pre-menopausal women who will not receive any chemoprevention drug (control)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Breast Density | up to 18 months
  Breast Density

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O' Sullivan, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (4):
- United States (4):
  - Pacific Breast Care Medical Clinic, Costa Mesa, California
  - Beckman Laser Institute Medical Clinic, Irvine, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Helen Diller Family Comprehensive Cancer Center/ UCSF, San Francisco, California